CLINICAL TRIAL: NCT02605889
Title: Acupuncture in the Treatment of Diabetes Mellitus Supplemental Type II : Applied Clinical Intervention by Nurses Acupuncturists
Brief Title: Acupuncture in the Complementary Treatment of Diabetes Mellitus Type II
Acronym: ACT-DM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: NEIDE APARECIDA TITONELLI ALVIM (Other)
Responsible Party: Sponsor-Investigator, NEIDE APARECIDA TITONELLI ALVIM, Phd Nursing, Universidade Federal do Rio de Janeiro
Organization: Universidade Federal do Rio de Janeiro (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 772.509
Record Dates: First submitted 2015-11-09; First posted 2015-11-16 (Estimated); Last update posted 2015-11-16 (Estimated); Status verified 2015-11

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A (Experimental): Laser acupuncture
  Interventions: Other: Laser acupuncture
- Group B (Sham Comparator): Simulation Laser acupuncture
  Interventions: Other: Laser acupuncture

INTERVENTIONS:
Other: Laser acupuncture — Laser acupuncture

SUMMARY:
This is a randomized clinical research, with triple blinded multicenter involving the Federal University of Rio de Janeiro, through the School of Nursing Anna Nery, as a proponent and research coordinator; and as a collaborative educational institutions, the Federal University of Espirito Santo, represented by the Department of Nursing; and the Higher School of Sciences of the Santa Casa de Misericordia de Vitoria, through the Master's Programme in Public Policy and Local Development.

As Research, the study covers health units of the Municipal Family Health Maricá / Rio de Janeiro, the Municipal Victoria Health / Holy Spirit, beyond the scope of Integrated Project Research-Service (PIPA), linked to Nursing Anna Nery / Federal University of Rio de Janeiro.

The object of investigation is the effectiveness of acupuncture in nursing care in complementary treatment of adult patients Diabetes Mellitus type II.

DETAILED DESCRIPTION:
This study has the general objective to evaluate the effectiveness of acupuncture as a complementary treatment to medication used in patients with diabetes mellitus type II, based on the nursing diagnoses.

ELIGIBILITY:
Inclusion Criteria:

* Be in possession of Diabetes Mellitus Type II only
* It is undergoing treatment for at least 1 year properly prescribed (to be confirmed with the medication of revenue)
* Report difficulties in glycemic control, regular saving measures higher than recommended by the Brazilian Society of Diabetes (postprandial up to 180mg / dl)

Exclusion Criteria:

* Have a lower limb amputated or part of them (because of the location of the selected acupoints for the treatment protocol)
* Be insulin
* Being a smoker
* Be alcoholic
* Be in drug treatment for other diseases including obesity
* Be making specific diet for weight loss
* Practicing regular physical activity
* Be in possession of cancer
* Being pregnant

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2014-10; Primary Completion 2015-12 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
Improvement of blood postprandial glucose levels | six week

SECONDARY OUTCOMES:
Improvement of Nursing Diagnoses | six week

CONTACTS AND LOCATIONS:
Overall Officials: Neide Alvim, PhD, Principal Investigator — Universidade Federal do Rio de Janeiro
Locations (1):
- Claudia Dayube Pereira, Rio de Janeiro, Rio de Janeiro, Brazil